CLINICAL TRIAL: NCT04858607
Title: Humoral and Cellular Immune Response to COVID-19 Vaccines in Immunocompromised and Healthy Individuals - The CoVVac Study
Brief Title: Humoral and Cellular Immune Response to COVID-19 Vaccines in Immunocompromised and Healthy Individuals
Acronym: CoVVac
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: CoVVac
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2023-02-09 (Actual); Status verified 2023-02

CONDITIONS: Covid19; Immunosuppression
Keywords: Vaccination
MeSH Terms: conditions — COVID-19 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — All samples will be stored at the Biobank of the Medical University of Graz for further analysis.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Immunocompromised individuals: Patients with primary or secondary immunodeficiency planning on vaccination against SARS CoV-2 according to the Austrian vaccination plan.
  Interventions: Diagnostic Test: Blood sample; Diagnostic Test: Saliva sample
- Healthy individuals: Healthy people planning on vaccination against SARS CoV-2 according to the Austrian vaccination plan.
  Interventions: Diagnostic Test: Blood sample; Diagnostic Test: Saliva sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Serology, immune status, T cell immunity, and T cell aging.
Diagnostic Test: Saliva sample — Antibody tests

SUMMARY:
Currently, the efficacy of COVID-19 vaccination in immunodeficient patients is unknown. Here the investigators aim to evaluate the efficacy of COVID-19 vaccines in immunodeficient patients compared to healthy controls. The investigators will assess the humoral and cellular response to COVID-19 vaccination in these subjects in detail. Furthermore, factors associated with good response to vaccination will be identified. The results of this study will help to guide future recommendations on COVID-19 vaccination in this population.

DETAILED DESCRIPTION:
The total duration of the study is 38 months, starting in March 2021 with a recruiting period until 31. December 2021 and termination of all scheduled visits until 31 May 2024. Individuals having consented and fulfilling the inclusion and exclusion criteria are included in the trial. A baseline visit will take place up to 60 days before the planned date of vaccination according to the Austrian vaccination plan. Scheduled vaccination with any COVID-19 vaccine approved in Austria will allow recruitment. If appropriate pre-vaccine samples from study participants exist in the biobank of the Medical University of Graz, patients may also be included in the study after vaccination starting with visit 3. In this case the biomaterial available at the biobank will be used for the analyses planned on visit 1. The investigators will not influence the date of vaccination or the type of the vaccine used. After first vaccination a telephone visit (visit 2) will assess adverse events and schedule visit 3 at the appropriate time after the second vaccination. At visit 3 the patient's vaccination certificate will be checked to verify correct vaccination and document the type of vaccine received. Further visits (5-6) will be performed for up to two years after the second vaccination. This follow-up period will allow an assessment of the duration of the immune response. The data recorded directly on the Case Report Form (CRF) are considered to be source data. COVID-19 vaccination, COVID-19 infection, Vaccination history, Pregnancy test, Adverse Events, BMI (Body Mass Index), and Laboratory Specimen Collection are recorded directly on the CRF and therefore are considered to be source data. Data will be merged in an electronic database (RDA Research, Documentation & Analysis; Medical University of Graz, version 07.03.2019). Case Report Forms (CRFs) will be inspected in respect of their accuracy and completeness and compared to original data by the monitor.

ELIGIBILITY:
Inclusion Criteria:

1. Noninfectious immunocompetent participants (i.e., healthy participants) as determined by medical history and clinical judgement.

   or
2. Patients with primary immunodeficiencies or
3. Patients with B-cell depleting therapy due to autoimmune disease or
4. Patients with benign and malignant hematological diseases receiving specific Treatments with known immunosuppressive effects including cytotoxic agents, systemic corticosteroids, monoclonal antibodies and targeted therapies.

   or
5. Patients with active hematological diseases and secondary immunoglobulin deficiency (e.g. chronic lymphatic leukemia, MM) currently not receiving specific treatment.

   or
6. Patients >3 months but <12 months after autologous HSCT (hematopoietic stem cell transplantation).

   or
7. Patients >3 months but <12 months after allogeneic HSCT. or
8. Recipients of HSCT >12 months after allogeneic HSCT but under immunosuppressive therapy.

   or
9. Patients with chronic GvHD (graft-versus-host disease) and persistent immunodeficiency.

Exclusion Criteria:

Healthy participants

1. Presence of diseases or therapies that are likely to interfere with the immune response to vaccination.
2. Presence of a disease requiring change in therapy during 4 weeks before enrollment.
3. Any contraindications to the vaccine planned to receive as listed in the product characteristics.
4. Lack of willingness to undergo serial blood draws and attend follow-up appointments.
5. Women who are pregnant or breastfeeding.
6. Previous vaccination with any coronavirus vaccine.
7. Persons who are not willing to sign the informed consents (biobank informed consent and study specific informed consent).

Immunodeficient participants

1. Patients with hematological diseases within three months from B-cell-depleting immunotherapy (rituximab, ofatumumab, obinutuzumab, blinatumomab, CAR-T cells (Chimeric Antigen Receptor).
2. Patients with hematological malignancies in remission and >12 months after end of specific therapy.
3. Patients within three months from HSCT.
4. Any contraindications to the vaccine planned to receive as listed in the product characteristics.
5. Lack of willingness to undergo serial blood draws and attend follow-up appointments.
6. Women who are pregnant or breastfeeding.
7. Previous vaccination with any coronavirus vaccine (exception: if serum prior to vaccination is available from the biobank).
8. Patients who are not willing to sign the informed consents (biobank informed consent and study specific informed consent).

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Immunodeficient participants and immunocompetent participants (i.e., healthy participants)
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2021-04-19 (Actual); Primary Completion 2023-01-20 (Actual); Study Completion 2023-01-20 (Actual)

PRIMARY OUTCOMES:
The levels of anti-SARS-CoV-2 spike protein humoral immune response. | At day 21-28 after the second vaccination
  The levels of anti-SARS-CoV-2 (severe acute respiratory syndrome-Covid Virus) spike protein humoral immune response measured by SARS-CoV-2 antigen-binding Ig assay comparing immunocompromised patients to healthy controls.

SECONDARY OUTCOMES:
Seroconversion | 6, 12 and 24 months after vaccination.
  Change of Seroconversion measured by SARS-CoV-2 antigen-binding Ig assay 6, 12 and 24 months after vaccination.
Concentrations of recombinant S protein-binding IgG (immunoglobulin G) | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Change of Concentrations of recombinant S protein-binding IgG after second vaccination in comparison to response after first vaccination.
Concentrations of secretory and serum IgA in comparison to IgG and IgM (immunoglobulin M) | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Change of Concentrations of secretory and serum IgA in comparison to IgG and IgM after second vaccination in immunocompromised, in recovered individuals and in healthy controls.
IFNγ production of T cells | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Change of IFNγ (Interferone gamma) production of T cells after SARS-CoV-2 antigen exposure, measured by FACS (fluorescence-activated cell sorter) and ELISpot.
Cross-reactive antibodies predicting the response to COVID-19 vaccinations | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Identification of parameters predicting the response to COVID-19 vaccinations: prior CoV infection (cross-reactive antibodies). Evaluation of the influence of previous infections caused by endemic CoV (proven through cross-reactive antibodies) on the vaccine response in immunocompromised individuals and in COVID-19 recovered individuals compared to controls.
Quantitative immunoglobulins predicting the response to COVID-19 vaccinations | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Identification of parameters predicting the response to COVID-19 vaccinations: quantitative immunoglobulins.
B cell subsets predicting the response to COVID-19 vaccinations | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Identification of parameters predicting the response to COVID-19 vaccinations: B cell subsets.
T cell subsets predicting the response to COVID-19 vaccinations | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Identification of parameters predicting the response to COVID-19 vaccinations: T cell subsets.
T cell aging predicting the response to COVID-19 vaccinations | 60-0 days before first vaccination.
  Identification of parameters predicting the response to COVID-19 vaccinations: T cell aging (TCR diversity, telomere length, TREC levels).
Occurence of neutralizing antibodies by means of SARS-CoV-2 neutralizing assays. | At day 21-28 as well as 12 and 24 months after the second vaccination.
  Neutralizing capacity of antibodies in respect of different SARSCoV-2 variants.
Correlation of diet and body fat with seroconversion | At day 21-28 and 12 months after the second vaccination.
  Correlation of diet and body fat with seroconversion after second vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stradner, Prof., Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No